CLINICAL TRIAL: NCT00593801
Title: Multicentre, Blinded, Randomised, Controlled Study on the Efficacy and Safety of Early or Late Epoetin Beta Treatment in Premature Infants (500- 999g Birth Weight)for Prevention or Treatment of Anaemia of Prematurity
Brief Title: Erythropoietin Treatment in Extremely Low Birth Weight Infants
Acronym: EPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Hoffmann-La Roche (Industry); University Hospital Tuebingen (Other); Children's Hospital at the Bult Hannover, Germany (Unknown); University Hospital, Aachen (Other); University of Zurich (Other); Children's Hospital Koeln, Germany (Unknown); Université Catholique de Louvain (Other); Children's Hospital Dortmund, Germany (Unknown); Hopital Antoine Beclere (Other); Hôpital Edouard Herriot (Other); Olga Hospital Stuttgart, Germany (Unknown); University Hospital, Strasbourg, France (Other)
Responsible Party: Prof. Dr. Michael Obladen, former Head of the Dpt. of Neonatology Charité Berlin, University Medicine Berlin, Charité
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12008; Hoffmann- La Roche,MF 4481
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Infant, Low Birth Weight; Anemia
Keywords: extremely low birth weight infants; transfusion need; erythropoietin; trace elements; antioxidant enzymes; reduction of the transfusion need by EPO treatment; trace elements and antioxidant enzymes in blood
MeSH Terms: conditions — Anemia | interventions — epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2: late rhEPO (Active Comparator): late EPO treatment from the fourth week for 6 weeks
  Interventions: Drug: epoetin beta
- 3: no EPO (No Intervention): control group, no EPO treatment
- 1: early rhEPO (Active Comparator): early rhEPO treatment from the first week until 9 weeks
  Interventions: Drug: epoetin beta

INTERVENTIONS:
Drug: epoetin beta — 250 IU/kg/week rhEPO treatment subcutaneously 3 times a week from the first week for 9 weeks, all infants received enteral iron 3-9 mg/kg/day
  Arms: 1: early rhEPO
Drug: epoetin beta — 250 IU/kg/week subcutaneously 3 times a week, from the fourth week for 6 weeks, all infants received enteral iron 3-9 mg/kg/day
  Arms: 2: late rhEPO

SUMMARY:
Objective: To investigate whether recombinant EPO reduces the need for transfusion in extremely low birth weight (ELBW) infants and to determine the optimal time for treatment.

The concentrations of trace elements and of antioxidant enzymes were investigated in all patients, too.

Study population: 219 patient randomized into 3 groups

DETAILED DESCRIPTION:
Methods: Blinded , multicenter trial, ELBW infants were randomized on day 3 to one of 3 groups: early EPO group (rhEPO from the first week for 9 weeks , n= 74), late rhEPO group (rhWEPO from the fourth week for 6 weeks, n=74), or control group (no rhEPO, n= 71). All infants received enteral iron (3-9 mg/kg/day) from the first week. The rhEPO ß dose was 750 IU/kg/week. Success was defined as no transfusion and hematocrit levels never below 30%.

The concentrations of trace elements and of antioxidant enzymes were investigated in all patients, too. Clinical and nutritional data were recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Extremely low birth weight infants

Exclusion Criteria:

* Cyanotic heart disease
* Major congenital malformation requiring surgery
* Gestational age > 30 weeks
* Administration of an investigational drug during pregnancy
* Lack of parental consent

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 1998-05; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
transfusion need | 9 weeks

SECONDARY OUTCOMES:
concentrations of trace elements and antioxidant enzymes in the blood | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Obladen, Prof.Dr., Principal Investigator — Charité Berlin, University Medicine
Locations (1):
- Dept of Neonatolgy Charité University Medicine Berlin, Berlin, State of Berlin, Germany